CLINICAL TRIAL: NCT06496308
Title: A Multicenter, Open-label, Randomized Controlled Study of Orelabrutinib in Combination With Bendamustine and Rituximab Versus Bendamustine and Rituximab in the Treatment of Transplant-Ineligible, Intermediate- to High-Risk Mantle Cell Lymphoma (MCL)
Brief Title: Bendamustine and Rituximab With or Without Orelabrutinib in MCL Treatment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: The Third Xiangya Hospital of Central South University (Other); Anhui Provincial Cancer Hospital (Other); Fujian Medical University Union Hospital (Other); Yantai Yuhuangding Hospital (Other); Huadong Hospital Affiliated with Fudan University, Shanghai (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Jiangxi Provincial Cancer Hospital (Other); Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORDER
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Mantle Cell Lymphoma (MCL)
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — orelabrutinib; Bendamustine Hydrochloride; Rituximab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Orelabrutinib + Bendamustine + Rituximab (OBR) (Experimental): In induction phase, patients will be randomized in two groups, one is OBR and another is BR. Patients in OBR group will receive rituximab 375 mg/m² IV on day 1, bendamustine 90 mg/m² IV on day 1 and 2, and orelabrutinib 150mg/day PO once daily, every 28 day per cycle for 6 cycles.
  Interventions: Drug: Orelabrutinib; Drug: Bendamustine; Drug: Rituximab
- Bendamustine + Rituximab (BR) (Placebo Comparator): In induction phase, patients will be randomized in two groups, one is OBR and another is BR. Patients in BR group will receive rituximab 375 mg/m² IV on day 1, bendamustine 90 mg/m² IV on day 1 and 2, every 28 day per cycle for 6 cycles.
  Interventions: Drug: Bendamustine; Drug: Rituximab
- Orelabrutinib + Venetoclax (OV) (Other): In maintanance phase, patients will receive different medical regimen according to their TP53 mutation and blastic and pleomorphic variants status. Patients with TP53 mutation or blastic and/or pleomorphic variant will receive orelabrutinib 150mg/day PO once daily and venetoclax for up to 2 years, the dosing of Venetoclax is escalated gradually to reach a target dose of 400 mg.
  Interventions: Drug: Orelabrutinib; Drug: Venetoclax
- Orelabrutinib (O) (Other): In maintanance phase, patients will receive different medical regimen according to their TP53 mutation and blastic and pleomorphic variants status. Patients without TP53 mutation or blastic and/or pleomorphic variant will receive orelabrutinib 150mg/day PO once daily for up to 2 years.
  Interventions: Drug: Orelabrutinib

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib PO will be administered as per the schedule specified in the respective arm.
  Arms: Orelabrutinib (O); Orelabrutinib + Bendamustine + Rituximab (OBR); Orelabrutinib + Venetoclax (OV)
Drug: Bendamustine — Bendamustine IV will be administered as per the schedule specified in the respective arm.
  Arms: Bendamustine + Rituximab (BR); Orelabrutinib + Bendamustine + Rituximab (OBR)
Drug: Rituximab — Rituximab IV will be administered as per the schedule specified in the respective arm.
  Arms: Bendamustine + Rituximab (BR); Orelabrutinib + Bendamustine + Rituximab (OBR)
Drug: Venetoclax — Venetoclax PO will be administered as per the schedule specified in the respective arm.
  Arms: Orelabrutinib + Venetoclax (OV)

SUMMARY:
This multicenter, open-label, randomized controlled trial aims to evaluate the efficacy and safety of Orelabrutinib in combination with Bendamustine and Rituximab (OBR) versus Bendamustine and Rituximab (BR) in patients with intermediate- to high-risk mantle cell lymphoma (MCL) who are ineligible for transplantation. The primary objective is to assess the complete response (CR) rate during the induction phase, with secondary objectives including progression-free survival (PFS), overall survival (OS), objective response rate (ORR), and safety. Exploratory analysis will investigate the correlation between tumor biomarkers and treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MCL (mantle cell lymphoma) through flow cytometry or histopathology, and has not received prior treatment.
* Age > 18 years of age, both genders are eligible.
* Ann Arbor stage II-IV; for stage II subjects, those who require systemic therapy based on the investigator's judgment are eligible.
* At least one measurable lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
* Any one of the following high-risk factors is present: MIPI score of 4-11, Ki67 > 50%, TP53 abnormality, blastic or pleomorphic variation.
* Patients who are not suitable candidates for autologous hematopoietic stem cell transplantation.
* Laboratory tests (blood routine, liver and kidney function) meet the following requirements: a) Blood routine: White blood cell count ≥3.0×10^9/L, absolute neutrophil count ≥1.5×10^9/L, hemoglobin ≥90g/L, platelet count ≥75×10^9/L. b) Liver function: Transaminases ≤2.5 times the upper limit of normal, bilirubin ≤1.5 times the upper limit of normal. c) Serum creatinine 44-133 mmol/L.
* The investigator judges that the subject's life expectancy is greater than 12 weeks from the time of screening.
* Willing and able to participate in all required assessments and procedures of the study protocol.

Exclusion Criteria:

* Patients who have previously received treatment with BTK inhibitors.
* Patients with severe complications or serious infections.
* Patients with uncontrolled cardiovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases, etc.
* Patients with active infections requiring systemic treatment, including bacterial, fungal, and viral infections.
* HIV-infected individuals.
* Patients with mental disorders or those who are known or suspected to be unable to fully comply with the study protocol.
* Patients whom the investigator judges to have other conditions that make them unsuitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2027-07-10 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | End of induction treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=28 days]
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Overall Response Rate | End of induction treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=28 days]
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Progression-free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No